CLINICAL TRIAL: NCT02084966
Title: Non-Invasive Evaluation of Transplant Kidney Using OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01DK094877 (NIH)
Record Dates: First submitted 2014-03-06; First posted 2014-03-12 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney; Transplantation; Imaging; Renal function; Optical Coherence Tomography
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCT Imaging (Experimental): OCT imaging of the kidneys prior to and following their transplant
  Interventions: Procedure: Procedure/Surgery: Transplantation: OCT of Kidney Transplant

INTERVENTIONS:
Procedure: Procedure/Surgery: Transplantation: OCT of Kidney Transplant — Device: Optical Coherence Tomography of Kidney Transplant

SUMMARY:
Optical coherence tomography (OCT) is a rapidly emerging imaging modality that can function as a type of "optical biopsy", providing non-invasive cross-sectional images of tissue architectural morphology in situ and in real-time. This proposal will demonstrate that OCT has the ability to provide novel and valuable histopathological information regarding donor kidneys that can be used to predict post-transplant renal function. These investigations will result in a major breakthrough in increasing the number of healthy kidneys available for transplantation by making the most efficient use of available donor kidneys, eliminating the possible use of bad donor kidneys, providing an accurate measure of expected post-transplant renal function, and allowing better distinction between post-transplant immunological rejection and ischemic-induced acute renal failure.

DETAILED DESCRIPTION:
What will be assessed: Kidney pathology will be assessed. Specifically, optical coherence tomography (OCT) will be used to observe the pathology of the kidney uriniferous tubules. The proximal convoluted tubules that make up most of the kidney uriniferous tubules and parenchyma in the outer cortex of the kidney (i.e., the portion of the kidney subjacent to the outer kidney capsule) are sensitive indicators of damage to the kidneys. When damaged due to ischemia (i.e., a lack of blood flow), these tubules swell and cellular debris is released into the lumens of these tubules.

Why is this data important: Damage to the kidney proximal tubules, known as acute tubular necrosis (ATN), is the most common cause of poor post-transplant kidney function following transplant. It has been shown that determining the extent of ATN is a good indicator of post-transplant renal function.

How will the data be collected: The histopathology describe above (i.e., the pathology of the kidney tubules) will be collected using optical coherence tomography (OCT). OCT is a rapidly emerging imaging modality that can function as a type of "optical biopsy", providing non-invasive cross-sectional images of tissue architectural pathology in situ and in real-time. OCT is similar to ultrasound, but uses light waves instead of sound waves to obtain high-resolution imaging. The ability of OCT of obtain high-resolution images is necessary in order to observe the pathological changes describe above (i.e., damage to the kidney tubules). Algorithms will be developed as a result of this investigation in order to assist in the prediction of ATN and post-transplant kidney function.

What factors will be measured to determine post-transplant kidney function: The factors that will be used to measure post-transplant renal function include serum creatinine, BUN and glomerular filtration rates (GFR). This data will be collected by examining the surgical and laboratory reports for each patient. The data will be collected daily for the first two weeks following transplant and biweekly for the next six months following transplant. Six months following transplant, this data will be collected every 3 months until conclusion of study (i.e., 4 years). The patient data will be stored on password-protected files on a password-protected computer. The data will be available only to the principal investigator and the co-investigators in this study. A nephrologist fellow who will report directly to the principal investigator will collect the data. The principal investigator will verify data accuracy and protocol compliance. A biostatistician who will be blinded as to patient identity will independently analyze the data. If the data is published, only the parameters listed above and related to post-transplant renal function will be reported. No names will be associated with publication of the collected kidney transplant data. The principal investigator and the biostatistician will monitor this data and any indications of potential harm to the patient will be reported immediately to the Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria: Undergoing Kidney Transplant -

Exclusion Criteria: None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2014-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Non-Invasive Evaluation of Transplant Kidney using OCT | Up to 4 years
  The outcome from these studies is to show significance differences in the donor kidneys of the three patient populations (i.e., immediate graft function, slow graft function and delayed graft function) using OCT imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States